CLINICAL TRIAL: NCT06666114
Title: Psoriatic Disease and Related Manifestations; Real World Evidence in Brazilian Secukinumab Environment
Status: Completed | Type: Observational
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CAIN457FBR04
Record Dates: First submitted 2024-10-29; First posted 2024-10-30 (Actual); Last update posted 2024-10-30 (Actual); Status verified 2024-10

CONDITIONS: Psoriasis (PsO); Psoriatic Arthritis (PsA)
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective

SUMMARY:
This was a retrospective observational study that relied on data extracted from patient chart review at the participating sites. At least 12 months of patient data was verified, comprising at least 6 months (pre-period) and 6 months (post-period) after secukinumab initiation (index date). All data extracted from patient charts was entered into an electronic case report form (eCRF), specifically designed to capture all variables needed for the study data analysis.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients aged ≥18 years at index date.
* Patients with PsO diagnosed with PsA (concomitant or sequentially), either by a rheumatologist or dermatologist, at least 6 months prior to initiation of secukinumab treatment.
* Continuously treated with secukinumab for at least 24 weeks (6 months) after index date.
* Medical history available from at least the one-year study period (at least 6 months previous to the start of secukinumab treatment and at least 6 months after).

Exclusion Criteria:

* Patients who interrupted secukinumab treatment for 3 or more months during the 6-month period (post-period) for any cause.
* Patients known to be participating in an interventional study at any point of the one-year study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This was a retrospective, noninterventional cohort study.
Sampling Method: Non-Probability Sample
Enrollment: 232 (Actual)
Dates: Start 2021-08-03 (Actual); Primary Completion 2023-10-10 (Actual); Study Completion 2023-10-10 (Actual)

PRIMARY OUTCOMES:
Proportion of Patients With Disease-related Clinical Manifestations During 6 Months Before and 6 Months After Secukinumab Initiation | Up to 1 year
Proportion of Patients With Disease-related Clinical Manifestations During 6 Months Before Secukinumab Introduction Who Experienced Reduced or Eliminated Manifestations During 6 Months of Secukinumab Treatment | Up to 1 year
Proportion of Patients With Disease-related Clinical Manifestations During 6 Months Before Secukinumab Introduction Who Experienced Increased Clinical Manifestations During 6 Months of Secukinumab Treatment | Up to 1 year
Proportion of Patients With Disease-related Clinical Manifestations at the Time of Secukinumab Introduction Who Experienced Reduced or Eliminated Manifestations During 6 Months of Secukinumab Treatment | Up to 6 months
Proportion of Patients With Disease-related Clinical Manifestations at the Time of Secukinumab Introduction Who Experienced Increased Manifestations During 6 Months of Secukinumab Treatment | Up to 6 months

SECONDARY OUTCOMES:
Age | Baseline
Gender | Baseline
Ethnicity | Baseline
Time Since First PsA Symptoms | Baseline
Time Since First PsO Symptoms | Baseline
Proportion of Patients With Disease-related Clinical Manifestations at Diagnosis | Baseline
Proportion of Patients per Screening Tool Used for PsA and PsO Diagnosis | Up to 1 year
  PsA and PsO screening tools included Psoriasis Area and Severity Index (PASI), Body Surface Area (BSA), Dermatology Life Quality Index (DLQI), Disease activity in PsA (DAPSA), and Health Assessment Questionnaire Disability Index (HAQ-DI).
Psoriasis Area and Severity Index (PASI) | Up to 1 year
  PASI is a combined assessment of lesion severity and affected area into a single score: 0 (no disease) to 72 (maximal disease).
Body Surface Area (BSA) | Up to 1 year
Dermatology Life Quality Index (DLQI) | Up to 1 year
  The DLQI is a validated, 10-question, self-reported questionnaire to evaluate the patient's perception of the impact of skin disease on quality of life. The DLQI is rated on a 4-point scale (0 = not at all to 3 = very much). The highest possible total score for the DLQI is 30, and higher scores indicate more severe impact on quality of life.
Disease activity in PsA (DAPSA) | Up to 1 year
  The Disease Activity Index for Psoriatic Arthritis (DAPSA) is a tool used to measure PsA activity: remission (0-4); low disease activity (5-14); moderate disease activity (15-28); high disease activity (>28).
Health Assessment Questionnaire Disability Index (HAQ-DI) | Up to 1 year
  The HAQ-DI is a 20-question scale assessing functional ability. The final HAQ-DI score ranges from 0 (no problems functioning) to 3 (not able to function).
Proportion of Patients per Treatment History Prior to Secukinumab Initiation | Up to 6 months
Proportion of Patients per Line of treatment (LOT) of PsA/PsO-target Treatment Before Secukinumab Initiation | Up to 6 months
Proportion of Patients With Disease-related Clinical Manifestations per Biologic Naïve and Non-biologic Naïve Patients, Categorized by Disease Severity | Up to 6 months
Proportion of Patients With Concomitant Medications, per Category | Up to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (1):
- Novartis, São Paulo, Brazil